CLINICAL TRIAL: NCT06083480
Title: Reducing Perioperative Oxidative Stress to Prevent Postoperative Chronic Pain Following Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Stephen Bruehl, PhD, Professor of Anethesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 231668; 1R01AG085287-01 (NIH)
Record Dates: First submitted 2023-10-05; First posted 2023-10-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis, Knee; Total Knee Arthroplasty; Chronic Postsurgical Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, mixed between/within-subject longitudinal trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GlyNAC (combination of glycine and n-acetylcysteine) (Experimental): GlyNAC 200 mg/kg/day (100mg glycine and 100mg N-acetyl-cysteine) will be administered orally in two divided doses each day for four weeks prior to TKA and six weeks postoperatively. The preparation will be a commercially available product of 1:1 ratio of glycine and N-acetyl-cysteine.
  Interventions: Drug: GlyNAC (combination of glycine and n-acetylcysteine)
- Placebo (alanine) (Placebo Comparator): Placebo (alanine) 200 mg/kg/day will be administered orally in two divided doses each day for four weeks prior to TKA and six weeks postoperatively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GlyNAC (combination of glycine and n-acetylcysteine) — GlyNAC 200 mg/kg/day (100mg glycine and 100mg N-acetyl-cysteine) will be administered orally in two divided doses each day for four weeks prior to TKA and six weeks postoperatively. The preparation will be a commercially available product of 1:1 ratio of glycine and N-acetyl-cysteine.
  Other Names: GlyNAC
  Arms: GlyNAC (combination of glycine and n-acetylcysteine)
Drug: Placebo — Placebo (alanine) 200 mg/kg/day will be administered orally in two divided doses each day for four weeks prior to TKA and six weeks postoperatively.
  Arms: Placebo (alanine)

SUMMARY:
This is a prospective randomized controlled trial that will assess preoperative, perioperative, and long-term oxidative stress (OS); pain; and functional outcomes over a 12 month period and test the hypothesis that a potent antioxidant intervention (glycine + N-acetyl-cysteine(GlyNAC)) reduces oxidative stress and chronic post surgical pain (CPSP) in patients undergoing total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
One of the most common surgical procedures performed in older adults is total knee arthroplasty (TKA), with an estimated 1 million TKAs performed annually in the United States. TKA directly addresses the pathology underlying knee joint pain and mobility limitations resulting from osteoarthritis. For most patients, TKA is effective for pain reduction and increasing function. However, a subgroup of 15-20% of TKA patients report unsatisfactory long-term pain outcomes well after postsurgical healing has occurred despite technical success of the procedure. Chronic postsurgical pain (CPSP) following TKA has been reported to be worse than the preoperative pain in 7% of TKA patients at up to 4-years. A potential biological mechanism is perioperative oxidative stress (OS),

The proposed project seeks to confirm the mechanistic role of OS in post-TKA CPSP and test the hypothesis that a perioperative intervention to reduce OS may reduce risk for CPSP post-TKA. This is a prospective randomized controlled trial that will assess preoperative, perioperative, and long-term oxidative stress (OS); pain; and functional outcomes over a 12 month period and test the hypothesis that a potent antioxidant intervention (GlyNAC) reduces OS and CPSP in patients undergoing total knee arthroplasty (TKA).

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* Intact cognitive status and ability to provide informed consent (based on cognitive screening with the Mini Mental State Examination)
* Ability to read and write in English sufficiently to understand and complete study questionnaires
* Undergoing unilateral primary TKA
* Medical diagnosis of osteoarthritis
* Past 24 hour worst numeric rating scale (NRS) pain of at least 4/10.

Exclusion Criteria:

* Diagnosis of pre-existing neuropathy
* Untreated hypo/hyperthyroidism
* Untreated heart disease
* Alanine transaminase/aspartate transaminase >2x upper-limit of normal range
* serum creatinine >1.5 mg/dl
* Pregnancy
* Complex Regional Pain Syndrome (CRPS) diagnosis prior to undergoing TKA
* Presence of lower extremity vascular disease, inflammatory or autoimmune disorders, or malignancy
* Presence of current clinically significant chronic pain conditions outside of the lower extremity ( daily pain for >3 months and greater ≥3/10 in intensity or the focus of medical care)
* Presence of other medical conditions that in the opinion of the orthopedic surgeon co-investigators would make a patient's study participation unsafe

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) Rating of Worst Pain in the past 24 hours | Baseline to 6 months post TKA (approximately 7 months)
  Mean within participant changes in NRS intensity ratings of worst pain in past 24 hours of measurement at 6 months post TKA. The score is a rating of current acute pain using a 0-100 numeric rating scale (NRS) (0 = "no pain" and 100 = "worst possible pain").

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) Rating of Worst Pain in the past 24 hours | Baseline to 6 weeks and 12 months post TKA (13 months)
  Mean within participant changes in NRS intensity ratings of worst pain in past 24 hours of measurement. The score is a rating of current acute pain using a 0-100 numeric rating scale (NRS) (0 = "no pain" and 100 = "worst possible pain")
Numeric Rating Scale of Average Pain in the past 24 hours | Baseline to 6 weeks, 6 months and 12 months post TKA (13 months)
  Mean within participant changes in NRS intensity ratings of average pain in past 24 hours of measurement. The score is a rating of current acute pain using a 0-100 numeric rating scale (NRS) (0 = "no pain" and 100 = "worst possible pain").
Numeric Rating Scale of Least Pain in the past 24 hours | Baseline to 6 weeks, 6 months and 12 months post TKA (13 months)
  Mean within participant changes in NRS intensity ratings of least pain in past 24 hours of measurement. The score is a rating of current acute pain using a 0-100 numeric rating scale (NRS) (0 = "no pain" and 100 = "worst possible pain").
Mean change in McGill Pain Questionnaire-2 (MPQ-2) ratings of knee pain for average pain over past week of measurement. | Baseline to 6 weeks, 6 months and 12 months post TKA (13 months)
  Mean within participant changes in McGill Pain Questionnaire-2 (MPQ-2) ratings of knee pain for average pain over past week of measurement. The MPQ-2 score ranges from 0-10 where 0 represents no pain and 10 represents the most intense pain.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS-JR) | Baseline to 6 weeks, 6 months and 12 months post TKA (13 months)
  Mean within participant changes in KOOS-JR ratings to assess movement evoked pain and functional limitations. Scores range from 0 to 100 with a score of 0 indicating total knee disability and 100 indicating perfect knee health.
PROMIS Short Form V1.0 - Pain Interference 8a scale | Baseline to 6 weeks, 6 months and 12 months post TKA (13 months)
  Mean within participant changes in PROMIS Short Form V1.0 - Pain Interference 8a scale to assess pain-related life interference over the week preceding assessments. This is an 8 item questionnaire with scores ranging from 0-40. 0 indicates no pain interference and 40 indicates the highest level of pain interference.
Postsurgical Opioid Use (pill count) | Post-TKA discharge to 6 weeks, 6 months and 12 months post-TKA (12 months)]
  Number of prescribed opioid pills used since hospital discharge following TKA. This is based on a combination of prescribed postsurgical opioid amounts and number of refills recorded in the electronic health record combined with pill counts conducted at each in-person post-TKA follow-up assessment.
Postsurgical Opioid Use (days of opioid use in the past week) | 6 weeks, 6 months and 12 months post-TKA (12 months)
  Number of days opioids were used in the past week at each in-person post-TKA follow-up assessment.
F2-Isoprostane/Isofuran (IsoP/IsoF) levels | Baseline to 4 week pre-TKA assessment, and 6 weeks, 6 months and 12 months post TKA (13 months)
  Changes in mean IsoP/IsoF levels from initial pre-intervention baseline. This is a measure of oxidative stress and is a mechanistic marker of the effects of the study antioxidant intervention (GlyNAC).
Glutathione levels | Baseline to 4 week pre-TKA assessment, and 6 weeks, 6 months and 12 months post TKA (13 months)
  Changes in mean glutathione levels from initial pre-intervention baseline. This is a measure of antioxidant capacity and is a mechanistic marker of the effects of the study antioxidant intervention (GlyNAC).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bruehl, Ph.D., Principal Investigator — Vanderbilt University Medical Center; Frederic T Billings, IV, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Key data elements will be preserved in final analyzed form (e.g., combined OS outcomes [mean of the two OS assays above], summary scores on all measures). The study protocol, standardized data collection instruments, and data dictionary will be uploaded in the repository. to facilitate study interpretation. Shared data will be uploaded in SPSS format.
  Data from the project will be stored within the Open Science Framework (OSF) database. OSF provides a unique URL for all datasets which will be provided for those interested. OSF also includes an interface with a search engine for identify datasets by topic/keyword.
  The data will be made available in OSF upon publication of the project findings. The data will continue to be available indefinitely on OSF subject to any OSF limitations. The dataset will be de-identified, so there will be no privacy limitations. Data will be accessible after publication of project results so there will be no limits on re-use.
Supporting Information: Study Protocol
Time Frame: The data will be made available in OSF upon publication of the project findings.
Access Criteria: OSF provides a unique URL for all datasets which will be provided for those interested. OSF also includes an interface with a search engine for identify datasets by topic/keyword.